CLINICAL TRIAL: NCT02058615
Title: Living With Hope: Development and Feasibility Evaluation of a Transition Toolkit for Make Partners of Women With Breast Cancer
Brief Title: Feasibility Testing and Evaluation of an Online Toolkit for Male Spouses of Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Wendy Duggleby, Professor and Nursing Research Chair, Aging and Quality of Life, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25908
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Male caregivers; Breast cancer; Intervention; Online toolkit
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Male Spouse Transition Toolkit (Experimental): All participants in this group will be given access to the Male Spouse Transition Toolkit (MaTT). MaTT is a website based application that is designed to help male spouses of women with breast cancer to increase their awareness of the transitions and experiences they have as a husband and caregiver as well as to stay organized and seek help and resources as needed. To do so it consists of six sections: about me; common changes to expect; frequently asked questions; resources; calendar; and, important health information. These sections contain activities and exercises, as well as fillable templates (i.e., resources, calendar) that users can download at their convenience, from their home computer, tablet, or smart phone. They will be asked to use the MaTT for one month.
  Interventions: Behavioral: Male Spouse Transition Toolkit
- Usual Care (No Intervention): Participants in this group will not receive access to the Male Spouse Transition Toolkit, and thus will not receive an intervention. Data collection for outcome variables will be the same as the participants in the experimental arm.

INTERVENTIONS:
Behavioral: Male Spouse Transition Toolkit
  Arms: Male Spouse Transition Toolkit

SUMMARY:
Male partners of women with breast cancer experience distress, so we want to develop a way to support them so they, in turn, can care for their wives. The purpose is to pilot test an online male spouse transition toolkit (MaTT) that the research team has developed. The specific aims are to: a) evaluate the Toolkit for ease of use, acceptability, and feasibility, and; b) collect preliminary data to determine potential effectiveness of the Toolkit in increasing hope, general self-efficacy and quality of life, and its potential effectiveness in decreasing guilt scores for male partners of women with breast cancer (stages 1-3).

ELIGIBILITY:
Inclusion Criteria:

* male
* 18 years of age or older
* living with a spouse who has breast cancer (Stage 1, 2, or 3)
* English speaking.

Exclusion Criteria:

* persons who are non-autonomous adults
* cognitively impaired as determined by the Registered Nurse (RN) researcher
* unable to participate, in the opinion of the RN researcher
* non-English speaking
* does not have a spouse who is diagnosed with having breast cancer (State 1, 2, or 3)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Hope | Change from baseline at day 7, 14, 28, and 56
  Hope is measured by the Herth Hope Index (HHI). The Herth Hope Index is a 12 item (1-4 point) Likert scale that delineates three sub-scales of hope: a) temporarility and future, b) positive readiness and expectancy, and c) interconnectedness. The HHI has been found to take approximately 5 minutes to complete. Summative scores range from 12-48, with a higher score denoting greater hope. This scale has been found to be reliable (test-retest r=91, p<0.05) and valid (concurrent validity, r=84, p.,0.05; criterion, r=92, p,0.05; divergent, r=-0.73, p. 0.05).

SECONDARY OUTCOMES:
Quality of Life | Change from baseline at day 7, 14, 28 and 56
  Caregiver quality of life is measured by the Caregiver Quality of Life-Cancer (CQOL-C) scale. This scale was developed specifically for family caregivers of persons with cancer. It consists of 35 items using a five-point Likert-type scale. It has four sub-scales: burden (physical and emotional), disruptiveness, positive adaptation and financial concerns. Higher scores reflect higher quality of life. It can be completed in 10 minutes and is considered easy to use. Test-retest reliability was found to be r=0.95 with an internal consistency of r=0.91. it was chosen for this study because it is easy to use and was developed based on quality of life studies of caregivers of persons with cancer.

OTHER OUTCOMES:
General self-efficacy | change from baseline at day 7, 14, 28, and 56
  General Self-efficacy is measured using the General Self-Efficacy Scale (GSES). This 10 item (0-4) Likert type scale produces a total perceived self-efficacy score. Higher scores indicate a higher self-efficacy or the confidence of one's ability to deal with adverse situations. It has a maximum score of 40.
Caregiver guilt | change from baseline at day 7 , 14, 28, and 56
  Caregiver guilt is measured by the Caregiver Guilt Questionnaire. This 22 item scale measures guilt on a five-point Likert scale (0 "Never" to 4 "Always") with a total range between 0 and 88. A higher score indicates that the respondent experienced more feelings of guilt related to their care giving. Cronbach's alpha indicated excellent internal consistency at 0.926.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy D Duggleby, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada